CLINICAL TRIAL: NCT01470742
Title: A Randomized, Phase III, Multicenter Clinical Trial Comparing Capecitabine Plus Oxaliplatin (XELOX) and Capecitabine (X) as First-line Chemotherapy in Elderly Patients With Advanced Gastric Cancer
Brief Title: Trial Comparing Capecitabine Plus Oxaliplatin (XELOX) and Capecitabine (X) as First-line Chemotherapy in Elderly Patients With Advanced Gastric Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We stop because of problems such as insurance.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-04-118
Record Dates: First submitted 2011-11-07; First posted 2011-11-11 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XELODA (Active Comparator): Capecitabine 1000mg/m2 bid D1-14 every 3weeks
  Interventions: Drug: XELODA
- XELOX (Experimental): D1-14 Capecitabine 1000mg/m2 bid D1 Oxaliplatin 110mg/m2 + D5W 250ml over 2hr every 3weeks
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: XELOX — D1-14 Capecitabine 1000mg/m2 bid D1 Oxaliplatin 110mg/m2 + D5W 250ml over 2hr every 3weeks
  Arms: XELOX
Drug: XELODA — Capecitabine 1000mg/m2 bid D1-14 every 3weeks
  Arms: XELODA

SUMMARY:
The objective of the trial is to compare Overall survival between capecitabine plus oxaliplatin (XELOX) and capecitabine (X) as first-line chemotherapy in elderly patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70
2. Histologically or cytologically confirmed adenocarcinoma of the gastric
3. Advanced ,metastatic/recurrence gastric cancer
4. ECOG performance status of 0 to 2
5. Life expectancy≥3months
6. No history of any systemic anti-cancer chemotherapy (prior adjuvant chemoradiation or chemotherapy is allowed if the last date of drug administration is > 6months from the study entry date)
7. No history of radiation therapy about Target lesion. (Prior radiotherapy is permitted if it was not administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented, and provided it has been completed at least 4 weeks before randomization.
8. Adequate marrow functions (ANC ≥ 1,500/uL, PLT ≥100,000/uL)
9. Adequate renal functions (Creatinine ≤1.5mg/dL or Ccr ≥ 50ml/min)
10. Adequate hepatic functions ( bilirubin ≤ 2.0mg/dL, SGOT/SGPT < normal x 3)
11. provision of a signed written informed consent

Exclusion Criteria:

1. History of any medical or psychiatric condition
2. Active infections
3. Peripheral neuropathy with symptom(NCI-CTCAE ver. 3.0 >=Grade 1 )
4. symptomatic brain metastases
5. Double primary cancer (physician at the discretion of the other cancer cured the purpose of early cancer cases can be registered)
6. History of other malignancy except:

   Adequately treated non-melanomatous skin cancer or cervical carcinoma in situ
7. Known hypersensitivity to Fluoropyrimidines/platinum
8. Clinical significant cardiovascular disease (myocardial infarction, symptomatic coronary artery disease, congestive heart failure, severe arrhythmias)
9. Required immunosuppressive therapy(transplant patients, severe autoimmune disease)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival of XELOX(XELODA/oxaliplatin) vs X(XELODA) | 36months

SECONDARY OUTCOMES:
response rate | 36months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea